CLINICAL TRIAL: NCT04904965
Title: Frontal Electroencephalography of Neonatal Patients Under Sedation With Opioids and General Anesthesia With Propofol.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 200916011
Record Dates: First submitted 2021-05-12; First posted 2021-05-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia; Surgery; Neonate; Depth of Anesthesia
Keywords: propofol; neonate; deph of anesthesia; Electroencephalography; surgery

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 4 groups, of 5 patients each, to receive total intravenous anesthesia, with different propofol induction infusion rates: Group 1 (Propofol 2.0 mg/kg/hr); Group 2 (Propofol 4.0 mg/kg/hr); Group 3 (Propofol 6.0 mg/kg/hr); Group 4 (Propofol 8.0 mg/kg/hr).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Propofol Group 1 (Experimental): Patients will receive induction of anesthesia with Propofol at a rate of 2.0 mg/kg/hr.
  Interventions: Drug: Propofol Group 1
- Propofol Group 2 (Experimental): Patients will receive induction of anesthesia with Propofol at a rate of 4.0 mg/kg/hr.
  Interventions: Drug: Propofol Group 2
- Propofol Group 3 (Experimental): Patients will receive induction of anesthesia with Propofol at a rate of 6.0 mg/kg/hr.
  Interventions: Drug: Propofol Group 3
- Propofol Group 4 (Experimental): Patients will receive induction of anesthesia with Propofol at a rate of 8.0 mg/kg/hr.
  Interventions: Drug: Propofol Group 4

INTERVENTIONS:
Drug: Propofol Group 1 — Propofol 2.0 mg/kg/hr per 10 min
  Other Names: Group 1
  Arms: Propofol Group 1
Drug: Propofol Group 2 — Propofol 4.0 mg/kg/hr per 10 min
  Other Names: Group 2
  Arms: Propofol Group 2
Drug: Propofol Group 3 — Propofol 6.0 mg/kg/hr per 10 min
  Other Names: Group 3
  Arms: Propofol Group 3
Drug: Propofol Group 4 — Propofol 8.0 mg/kg/hr per 10 min
  Other Names: Group 4
  Arms: Propofol Group 4

SUMMARY:
Frequently, neonates hospitalized in neonatology units require anesthesia for surgery. The drugs used for this purpose are opioids and other anesthetics, such as propofol.

Currently, the administration of anesthesia is difficult in neonates due to the neurological immaturity of these patients, the scarcity of adequate pharmacological studies, the prolonged use of one or more sedatives prior to surgery and the limited usefulness of current anesthetic monitoring devices in this population.

Electroencephalography (EEG), which has allowed estimation of anesthetic depth in other populations, has been less explored in neonates. To date, there are no EEG markers, correlated with a given dose of anesthesia, that allow an adequate administration in this kind of patients. In this context, a better understanding of the anesthetic effect in the neonatal brain would allow defining characteristic EEG patterns, improving the estimation of anesthetic depth and anesthetic dosage in neonates.

DETAILED DESCRIPTION:
As a consequence of the cerebral immaturity of newborns (1,2), together with the fact that in the NICU it is common to find patients requiring surgery who are sedated with multiple drugs, it is necessary to define characteristic EEG patterns that allow estimation of the anesthetic depth and adequate dosage of anesthetics, avoiding the the risk of under- or overdosing of anesthetics (3).

The investigators will conduct an exploratory study. The aim of the study is to determine, by frontal electroencephalography, markers of brain electrical activity associated with the administration of propofol in term newborns requiring surgery in the NICU. A sample of 20 term neonatal patients admitted to the NICU UC with a diagnosis of surgical pathology will be included.

General objective:

To describe the characteristics of the frontal electroencephalographic pattern associated with increasing doses of propofol, in term neonates, requiring surgery in the NICU and its correlation with a clinical response, to the surgical stimulus.

Specific objectives:

* Identify the association between electroencephalographic parameters and different levels of sedation prior to surgery.
* To identify the association between electroencephalographic parameters and increasing doses (plasma concentration) of propofol administered in a previously sedated patient.
* To relate the clinical response observed to the surgical stimulus and increasing doses (plasma concentration) of propofol in a previously sedated patient (dose (concentration) - response curve).
* To describe the temporal profile of propofol anesthesia, based on the changes in electroencephalographic parameters observed over time, during the period of administration and suspension of the anesthetic.

On the scheduled day of surgery in the NICU and prior to anesthetic induction, in sedated and standardly monitored patients (ECG, SpO2, PAI, temperature, diuresis). A four-channel SedLine® monitor (Masimo Corporation, Irvine, CA, USA) will be used to monitor frontal brain electrical activity 10 minutes before the induction of anesthesia. At the end of this period, the level of sedation will be evaluated with the N-PASS clinical scale (4) and the types, doses and duration of sedative drugs administered up to that time will be recorded. Then, patients will be randomized into 4 groups, of 5 patients each, to receive manual total intravenous anesthesia, with different propofol infusion rates: Group 1, Propofol 2.0 mg/kg/hr; Group 2, Propofol 4.0 mg/kg/hr; Group 3, Propofol 6.0 mg/kg/hr; Group 4, Propofol 8.0 mg/kg/hrs. At 10 and 20 minutes after the start of the propofol infusion, arterial blood samples will be taken to determine the plasma concentration of propofol reached during the anesthetic induction. In case of hemodynamic alteration (heart rate and/or blood pressure drop by 20%) during the propofol infusion, a 25% decrease of the original dose will be performed. At the end of this period, surgery will be initiated. The hemodynamic and motor response to the surgical stimulus will be observed and recorded. If there is hemodynamic response (increase in heart rate and/or blood pressure by 20%) and/or motor response, after the surgical stimulus, fentanyl rescue 5 mcg/kg/iv will be administered. Subsequent anesthesia will be in the hands of the treating anesthesiologist in the doses and forms he/she deems convenient. Electroencephalographic tracing will be maintained continuously throughout the procedure (from 10 minutes before and up to 10 minutes after surgery). Changes and adjustments to the anesthesia and analgesia given, hemodynamic changes occurring during the procedure and anesthetic and surgical times will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (>37 weeks) admitted to the NICU
* Diagnosis of surgical pathology, non-neurological, to be resolved in the NICU, in the next hours or days.
* Need for continuous sedation-analgesia prior to surgery.

Exclusion criteria:

* Perinatal asphyxia
* Evidence of severe neurological injury.
* Suspected or diagnosed brain malformations
* Uncontrolled metabolic and hemodynamic instability at the time of surgery.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Electroencephalography monitoring slow bands | 10 minutes before the induction of anesthesia until 10 minutes after emergence of anesthesia, average of 2 hours
  Power of frequency slow bands, entropy and complexity measures.
Electroencephalography monitoring alpha bands | 10 minutes before the induction of anesthesia until 10 minutes after emergence of anesthesia, average of 2 hours
  Power of frequency alpha bands, entropy and complexity measures.
Electroencephalography monitoring Theta bands | 10 minutes before the induction of anesthesia until 10 minutes after emergence of anesthesia, average of 2 hours
  Power of frequency Theta bands, entropy and complexity measures.

SECONDARY OUTCOMES:
Arterial Pressure | From induction of anesthesia until surgery starts, average 20 minutes.
  By non invasive Arterial Pressure: Systolic Arterial Pressure in mmHg, diastolic Arterial Pressure in mmHg and Medium Arterial Pressure in mmHg, every 5 minutes.
Heart Rate | From induction of anesthesia until surgery starts, average 20 minutes.
  By EKG D-II, every 5 minutes.
Depth of anesthesia | before the induction of anesthesia until the surgery starts, every 10 minutes. An average of 30 minutes.
  Evaluated with N-PASS clinical scale. The N-PASS uses five criteria: crying/irritability, behavioral state, facial expression, extremity tone and vital signs. The scale has a range from 0 (normal) to -10 (sedated).
Propofol plasma concentration | from induction of anesthesia up to 20 minutes.
  Venous or arterial samples will be taken for propofol plasma concentration levels (ng/ml) at two times (10 minutes and 20 minutes from induction of anesthesia).
Motor response to surgical incision | at first surgical incision (average 1 minute).
  Presence of any body movement at the moment of the first surgical incision.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio C Ibacache, PhD, MD, Principal Investigator — Associate Professor
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre M, Lamblin MD, d'Allest AM, Curzi-Dascalova L, Moussalli-Salefranque F, S Nguyen The T, Vecchierini-Blineau MF, Wallois F, Walls-Esquivel E, Plouin P. Electroencephalography in premature and full-term infants. Developmental features and glossary. Neurophysiol Clin. 2010 May;40(2):59-124. doi: 10.1016/j.neucli.2010.02.002. Epub 2010 Mar 16. PMID 20510792
- [Background] Shany E, Berger I. Neonatal electroencephalography: review of a practical approach. J Child Neurol. 2011 Mar;26(3):341-55. doi: 10.1177/0883073810384866. PMID 21383227
- [Background] Anand KJ, Willson DF, Berger J, Harrison R, Meert KL, Zimmerman J, Carcillo J, Newth CJ, Prodhan P, Dean JM, Nicholson C; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Tolerance and withdrawal from prolonged opioid use in critically ill children. Pediatrics. 2010 May;125(5):e1208-25. doi: 10.1542/peds.2009-0489. Epub 2010 Apr 19. PMID 20403936
- [Background] Giordano V, Edobor J, Deindl P, Wildner B, Goeral K, Steinbauer P, Werther T, Berger A, Olischar M. Pain and Sedation Scales for Neonatal and Pediatric Patients in a Preverbal Stage of Development: A Systematic Review. JAMA Pediatr. 2019 Dec 1;173(12):1186-1197. doi: 10.1001/jamapediatrics.2019.3351. PMID 31609437
- [Derived] Boncompte G, Cortinez LI, Toso A, Giordano A, Cruzat F, Fuentes R, Pedemonte JC, Contreras V, Biggs D, Chiu E, Ibacache M. Differential effects of propofol anaesthesia across three amplitude-defined electroencephalographic states in sedated critically ill term neonates: An observational study. Eur J Anaesthesiol. 2025 Oct 1;42(10):889-898. doi: 10.1097/EJA.0000000000002208. Epub 2025 May 23. PMID 40420743